CLINICAL TRIAL: NCT00484224
Title: Audiological Disturbances in Vitiligo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: qwer1234-HMO-CTIL
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-05

CONDITIONS: Vitiligo; Hearing Loss
MeSH Terms: conditions — Vitiligo; Hearing Loss

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to determine wether vitiligo patients have more audiological abmnormalities, than the healthy population.

ELIGIBILITY:
Inclusion Criteria:

* vitligo patients under 50. healthy patients under 50 for control group

Exclusion Criteria:

* above age 50. systemic disease. exposure to loud noise in past. familial history of deafness use of autotoxuc drugs or steroids. autoimmune/metabolic/neurologic/vascular disease

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Arieh Ingber, Prof., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Aydogan K, Turan OF, Onart S, Karadogan SK, Tunali S. Audiological abnormalities in patients with vitiligo. Clin Exp Dermatol. 2006 Jan;31(1):110-3. doi: 10.1111/j.1365-2230.2005.02004.x. PMID 16309498